CLINICAL TRIAL: NCT06706154
Title: Determinants of Exercise Capacity in Kidney Transplant Recipients
Brief Title: Exercise Capacity in Kidney Transplant Recipients
Status: Recruiting | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Merve Firat, Assistant Professor, Hacettepe University
Other Study IDs: FTREK24/67
Record Dates: First submitted 2024-11-04; First posted 2024-11-26 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Renal Transplantation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Kidney transplant recipients

SUMMARY:
This study aimed to determine the determinants of 6 minute walk test distance in patients with kidney transplant recipients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with kidney transplantation
* At least 6 months after the kidney transplant
* Being aged 18-65
* Not having regular exercise habits
* Voluntary participation in the study

Exclusion Criteria:

* Having a musculoskeletal problem that may interfere with the tests
* Having neurological impairment
* Having chronic lung disease
* Having had any cardiovascular event in the last 6 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with kidney transplantation will be included.
Sampling Method: Non-Probability Sample
Enrollment: 27 (Estimated)
Dates: Start 2024-08-17 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Exercise capacity | 1st day
  Will be evaluated with 6 minute walk test. After the test, total walking distance will be recorded.
Respiratory function | 1st day
  FEV1, FVC, FEV1/FVC, PEF, FEF25-75 will be measured by lung function test.
Respiratory muscle strength | 1st day
  Maximal inspiratory pressure (MIP) and maximal expiratory pressure (MEP) will be measured using a mouth pressure device.
Musle function | 1st day
  Knee extensor and hand grip strength will be evaluated with a dynamometer.

SECONDARY OUTCOMES:
Physical activity | 1st day
  Physical activity level will be evaluated using International Physical Activity Questionnaire-Short form. This questionnaire lists activities and asks for estimates of the duration and frequency of each activity in the past week. The durations are multiplied by the MET value for each activity and the results for all items are summed to give an overall physical activity score.

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)